CLINICAL TRIAL: NCT04751968
Title: Building Resilience and Attachment in Vulnerable Adolescents (BRAVA): A Randomized Controlled Trial of a Brief Group Intervention for Adolescents With Mild to Moderate Suicidal Ideation and Their Caregivers
Brief Title: BRAVA: Building Resilience and Attachment in Vulnerable Adolescents
Acronym: BRAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Mach Gaensslen Foundation (Other); Children's Hospital of Eastern Ontario Research Institute (Other)
Responsible Party: Principal Investigator, Allison Kennedy, Principal Investigator, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1922_SI_Group
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation; Suicide and Self-harm
Keywords: Adolescent; Suicidal ideation; Group therapy; Crisis
MeSH Terms: conditions — Suicidal Ideation; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intervention (Experimental): The intervention will consist of 6 psycho-educational group sessions for caregivers and 6 psycho-educational group sessions for adolescents. Adolescent and caregiver sessions will be held separately and will focus on different issues. Adolescents are taught skills for coping and relating more effectively with others. Caregivers learn about adolescent development, effective parenting and the importance of connection. The groups consist of 6 stand-alone modules permitting rolling entry and prompt access. Youth and Caregivers will receive a weekly text message reminder of their exit assessment date/time, homework from that week's intervention group and crisis resources.
  Interventions: Other: Group Intervention
- Enhanced Treatment as Usual (Other): Youth and Caregivers will receive a weekly text message reminder of their exit assessment date/time, a mental health tip and crisis resources.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Other: Group Intervention — The intervention will consist of 6 psycho-educational group sessions for caregivers and 6 psycho-educational group sessions for adolescents. Adolescent and caregiver sessions will be held separately and will focus on different issues. Adolescents are taught skills for coping and relating more effectively with others. Caregivers learn about adolescent development, effective parenting and the importance of connection. The groups consist of 6 stand-alone modules permitting rolling entry and prompt access. Youth and Caregivers will receive a weekly text message reminder of their exit assessment date/time, homework from that week's intervention group and crisis resources.
  Arms: Group Intervention
Behavioral: Enhanced Treatment as Usual — Youth and Caregivers will receive a weekly text message reminder of their exit assessment date/time, a mental health tip and crisis resources.
  Arms: Enhanced Treatment as Usual

SUMMARY:
The prevalence of suicidal ideation (SI) among adolescents in North America is high, making it critical to develop evidence-based brief interventions for adolescents with SI that target healthy coping skills and relationships. BRAVA is a novel brief group intervention for adolescents with mild to moderate SI and their caregivers; youth are taught skills for coping and relating more effectively with others. Caregivers learn about adolescent development, effective parenting and the importance of connection. The goal of the randomized controlled trial is to assess the efficacy of a virtually-delivered, brief group intervention for adolescents with mild to moderate SI and their caregivers in reducing SI.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 13 years old to 17.5 years old
* Mild to moderate suicidal ideation (SI without plan or gesture; 1 on the HEADS-ED) (Cappelli, et al., 2012)
* Interested in study participation
* Access to an electronic device with internet and email capabilities, and a functioning camera and microphone

Exclusion Criteria:

* SI with plan or gesture (2 on HEADS ED; indicated plan or gesture)
* Comorbid disorders (psychosis, schizophrenia, developmental disabilities, major substance abuse, and severe eating disorders).
* Referring clinician has identified an externalizing disorder as a primary diagnosis or primary concern (e.g. Conduct Disorder)
* Currently participating in regular psychotherapy at least one time per week
* Currently under Children's Aid Society care
* Currently in the CHEO ED on a Form 1 or Form 2, or placed on a Section 17.
* Express difficulty with reading and writing

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation | 6 weeks
  Suicidal ideation will be measured using the Suicidal Ideation Questionnaire Junior (Reynolds, 1988). A decreased score in suicidal ideation over 6-weeks will indicate a positive outcome.

SECONDARY OUTCOMES:
Depression and Anxiety | 6 weeks
  We will be assessing youth depression and anxiety with the youth version of the Revised Child Anxiety and Depression Scale (Chorpita et al., 2000). A decreased score in depression and anxiety over 6-weeks will indicate a positive outcome.
Attachment | 6 weeks
  We will be assessing caregiver attachment with the adolescent version of the Adolescent Attachment Anxiety & Avoidance Inventory (Morretti & Obsuth, 2009). A decreased score in attachment between the adolescent and caregiver over 6-weeks will indicate a positive outcome.
Family Functioning | 6 weeks
  Family functioning using the Family Assessment Device (Epstein, Baldwin, & Bishop, 1983). A decreased score in family functioning over 6-weeks will indicate a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Kennedy, PhD, Principal Investigator — CHEO
Locations (1):
- CHEO, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Georgiades K, Boylan K, Duncan L, Wang L, Colman I, Rhodes AE, Bennett K, Comeau J, Manion I, Boyle MH; 2014 Ontario Child Health Study Team. Prevalence and Correlates of Youth Suicidal Ideation and Attempts: Evidence from the 2014 Ontario Child Health Study. Can J Psychiatry. 2019 Apr;64(4):265-274. doi: 10.1177/0706743719830031. PMID 30978144
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Reynolds, W. M. (1988). Suicidal Ideation Questionnaire Professional Manual (p. 47).
- [Background] Cloutier, P., Glennie, E., Kennedy, A., & Gray, C. (2009). Coping Behaviours and Non-Suicidal Self-Harm in Youth. In Canadian Psychological Association's 70th Annual Convention. Montreal, Quebec.
- [Background] Moretti MM, Obsuth I. Effectiveness of an attachment-focused manualized intervention for parents of teens at risk for aggressive behaviour: The Connect Program. J Adolesc. 2009 Dec;32(6):1347-57. doi: 10.1016/j.adolescence.2009.07.013. Epub 2009 Sep 18. PMID 19766302
- [Background] Epstein, N. B., Baldwin, L. M., & Bishop, D. S. (1983). The McMaster Family Assessment Device. Journal of Marital and Family Therapy, 9(2), 171-180.
- [Background] Cappelli M, Gray C, Zemek R, Cloutier P, Kennedy A, Glennie E, Doucet G, Lyons JS. The HEADS-ED: a rapid mental health screening tool for pediatric patients in the emergency department. Pediatrics. 2012 Aug;130(2):e321-7. doi: 10.1542/peds.2011-3798. Epub 2012 Jul 23. PMID 22826567
- [Derived] Kennedy A, Gray C, Sheridan N, Dunn L, Stewart J, Drouin S, Elliott H, Adeponle A, Barrowman N, Sucha E, Cappelli M, Norris ML, Jabbour M, Cloutier P. BRAVA: A randomized controlled trial of a brief group intervention for youth with suicidal ideation and their caregivers. Child Adolesc Psychiatry Ment Health. 2025 Jul 16;19(1):78. doi: 10.1186/s13034-025-00941-1. PMID 40671103
- See also: CHEO Research Institute — http://www.cheoresearch.ca